CLINICAL TRIAL: NCT06961318
Title: Arthroscopic Treatment of Rotator Cuff Tears
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20250255; BYSYDL2024014 (Other Grant/Funding Number: Peking University Third Hospital)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff
Keywords: Rotator cuff tear; arthroscopy; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Single Row Repair: Single Row Repair
- Double Row Repair: Double Row Repair
- M Type Repair: M Type Repair

SUMMARY:
Rotator cuff tears are the primary cause of shoulder pain and functional impairment, accounting for 50% to 85% of shoulder disorders. With the acceleration of population aging in China and the increasing demand for sports brought about by the improvement of economic standards, rotator cuff tears have gradually become a significant social health problem that cannot be ignored. Currently, arthroscopic rotator cuff repair is the standard treatment for rotator cuff tears. However, studies have shown that the average re-tear rate after rotator cuff repair surgery is 26.6%, which can be as high as 95% for massive rotator cuff tears. Therefore, how to prevent the occurrence of re-tears after arthroscopic rotator cuff repair and improve surgical outcomes has become a hot spot for research in the field of shoulder arthroscopy. Based on previous clinical experience, our team developed an M-shaped suture technique for arthroscopic rotator cuff repair. Clinical observations have shown that the re-tear rate at one-year post-surgery is 8%, which is significantly lower than what has been reported in the literature. However, there is currently a lack of comparative studies on the efficacy of this technique versus traditional single-row and double-row suture techniques. Moreover, the current research evidence on the prognostic factors affecting rotator cuff repair surgery is conflicting, and there is still a lack of high-quality cohort studies to screen for risk factors for poor prognosis. This project aims to establish a high-quality ambispective cohort for minimally invasive arthroscopic surgery for rotator cuff tears, to compare the clinical efficacy of the M-shaped suture technique with traditional techniques, and to identify risk factors related to the prognosis after rotator cuff repair surgery. This will provide high-quality, real-world evidence to optimize the new suture technique and develop a clinical prediction model for re-tears after rotator cuff suture repair. In the long term, the project will conduct embedded intervention studies to address modifiable risk factors (including lifestyle interventions and optimization of rehabilitation protocols) and verify whether these interventions can enhance prognostic outcomes, so as to better develop a more scientific and rational management and treatment plan for patients with rotator cuff tears. We aim to address the challenge of low tendon-bone healing rates and high re-tear rates in rotator cuff repair surgery, and provide reliable, effective, and cost-effective treatment options for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Primary arthroscopic rotator cuff repair
* Full-thickness rotator cuff tear confirmed by clinical examination and magnetic resonance imaging (MRI)
* Patient has signed the informed consent form
* Patient is willing and able to participate in follow-up and evaluation procedures

Exclusion Criteria:

* Partial rotator cuff tear or irreparable massive tear
* Concurrent shoulder pathologies other than rotator cuff injury, such as frozen shoulder or shoulder instability
* History of significant trauma to the ipsilateral shoulder
* History of previous surgery on the ipsilateral shoulder
* Presence of severe systemic diseases, such as tumors or severe dysfunction of internal organs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary arthroscopic rotator cuff repair
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Retear | Post-op 3 months, 1 year, 2 years
  Sugaya IV & V on MRI

SECONDARY OUTCOMES:
VAS-pain | Baseline, Post-op 3 months, 1 year, 2 years
  VAS-pain
ASES shoulder score | Baseline, Post-op 3 months, 1 year, 2 years
  ASES shoulder score
WORC | Baseline, Post-op 3 months, 1 year, 2 years
  WORC
EQ-5D | Baseline, Post-op 3 months, 1 year, 2 years
  EQ-5D
Constant-Murley shoulder score | Baseline, Post-op 3 months, 1 year, 2 years
  Constant-Murley shoulder score
Range of Motion | Baseline, Post-op 3 months, 1 year, 2 years
  Range of Motion

OTHER OUTCOMES:
Complications | Baseline, Post-op 3 months, 1 year, 2 years
  Hematoma, nerve injury, infection, anchor pull-out

CONTACTS AND LOCATIONS:
Overall Officials: Zhenxing Shao, MD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No